CLINICAL TRIAL: NCT00634842
Title: Effect of Two Different Fasting Blood Glucose Titration Targets in Glucose Control in Patients With Type 2 Diabetes Using Insulin Detemir Once Daily in Combination With 1-3 Oral Agents
Brief Title: Effect of Two Different Fasting Blood Glucose Targets on Glucose Control in Patients With Type 2 Diabetes Using Insulin Detemir Once Daily
Acronym: TITRATE™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-3502
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FPG 70-90 mg/dL (Experimental): Aggressive FPG (fasting plasma glucose) titration target range group
  Interventions: Drug: insulin detemir
- FPG 80-110 mg/dL (Experimental): Conventional FPG (fasting plasma glucose) titration target range group
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target dose titration scheme, s.c. injection, once daily. Fasting plasma glucose (FPG) titration target range of 70-90 mg/dL
  Arms: FPG 70-90 mg/dL
Drug: insulin detemir — Treat-to-target dose titration scheme, s.c. injection, once daily. Fasting plasma glucose (FPG) titration target range of 80-110 mg/dL
  Arms: FPG 80-110 mg/dL

SUMMARY:
This trial is conducted in the United States of America. The aim of this trial is to explore how different fasting blood glucose targets affect glucose control in patients with type 2 diabetes, when patients are empowered to do dose adjustments themselves.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* 1-3 oral treatments
* Insulin naive
* BMI (Body Mass Index) less than or equal to 45

Exclusion Criteria:

* Pregnancy
* Retinopathy
* Cardiac disease
* Uncontrolled hypertension
* Recurrent hypoglycaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (61):
- United States (58):
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Scottsdale, Arizona
  - Novo Nordisk Investigational Site, Searcy, Arkansas
  - Novo Nordisk Investigational Site, Artesia, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Parker, Colorado
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Prospect, Connecticut
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Terre Haute, Indiana
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Pikesville, Maryland
  - Novo Nordisk Investigational Site, Saint Paul, Minnesota
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Camden, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Shelby, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Taylors, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, Odessa, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Puerto Rico (3):
  - Novo Nordisk Investigational Site, Caguas
  - Novo Nordisk Investigational Site, San Juan
  - Novo Nordisk Investigational Site, Trujillo Alto

REFERENCES:
- [Result] Blonde L, Merilainen M, Karwe V, Raskin P; TITRATE Study Group. Patient-directed titration for achieving glycaemic goals using a once-daily basal insulin analogue: an assessment of two different fasting plasma glucose targets - the TITRATE study. Diabetes Obes Metab. 2009 Jun;11(6):623-31. doi: 10.1111/j.1463-1326.2009.01060.x. PMID 19515182
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 69 sites in the United States of America (USA).
Pre-assignment Details: Subjects were randomised 1:1 to 2 FPG (fasting plasma glucose) titration targets. Insulin doses were self-titrated every three days based on self-measured FPG levels as follows: -3 units if FPG was below the lower limit of the target range, no change if FPG was within target range, and +3 units if FPG was above the upper limit of the target range.
Period: Overall Study
Arm/Group | FPG 70-90 mg/dL | FPG 80-110 mg/dL
Started | 122 | 122
Completed | 107 | 104
Not Completed | 15 | 18
Not completed — Adverse Event | 2 | 3
Not completed — Protocol Violation | 8 | 4
Not completed — Move to another state | 1 | 0
Not completed — Inclusion criteria were not met | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lack of time and intolerance to drug | 0 | 1
Not completed — Discontinued due to injection | 0 | 2
Not completed — No need of study drug to treat diabetes | 0 | 1
Not completed — No wish to keep taking Avandia | 0 | 1
Not completed — Subject off study drug for too long | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FPG 70-90 mg/dL | FPG 80-110 mg/dL | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.4) | 57.2 (10.6) | 56.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 44 | 98
  Male | 68 | 78 | 146
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Level of fasting plasma glucose (FPG) measured at baseline
  mg/dL | 164.0 (43.1) | 163.1 (40.4) | 163.5 (41.7)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage] — Level of glycosylated haemoglobin (HbA1c) measured at baseline
  percentage | 8.0 (0.6) | 7.9 (0.6) | 8.0 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Glycosylated Haemoglobin A1c (HbA1c) Less Than 7%
Description: Percentage (%) of subjects reaching glycosylated haemoglobin A1c (HbA1c) less than 7% measured after 20 weeks of treatment
Time Frame: week 20
Population: The intent-to-treat (ITT) population with non-missing HbA1c values at end of study, LOCF (last observation carried forward)
Measure: Number; unit: percentage of participants
Arm/Group | FPG 70-90 mg/dL | FPG 80-110 mg/dL
Number analyzed (Participants) | 112 | 112
percentage of participants | 64.3 | 54.5
Statistical Analysis 1: Comparison: FPG 70-90 mg/dL vs FPG 80-110 mg/dL; To show non-inferiority for the primary endpoint, 100 subjects per group provides 80% power to show that the 95% CI for the difference of proportions between treatments is within the 20% margin under the assumption of equality of proportions. It is also sufficient to show superiority under the assumption that the first proportion is greater than the second by at least 20%. With a predicted withdrawal rate of 15%, 236 subjects were needed based on a treatment ratio of 1:1 for the two treatments; Test type: Non-Inferiority or Equivalence — The primary hypothesis was that there would be no difference in efficacy as measured by the proportion of subjects reaching HbA1c level < 7% between the two FPG titration arms (70-90 mg/dL and 80-110 mg/dL, respectively) with a non-inferiority margin of 20%. If non-inferiority of the 70-90mg/dL arm was established, superiority was to be tested using a Logistic regression model with baseline HbA1c as a covariate. Superiority was to be concluded if the odds ratio was significantly greater than 1; p = 0.0411, Test for Difference in Proportions; Odds Ratio (OR) = 1.86, 95% CI [1.03 to 3.37]

2. Secondary Outcome: Percentage of Participants Achieving Glycosylated Haemoglobin A1c (HbA1c) Less Than or Equal to 6.5%
Description: Percentage (%) of participants reaching glycosylated haemoglobin A1c (HbA1c) less than or equal to 6.5% measured after 20 weeks of treatment
Time Frame: week 20
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | FPG 70-90 mg/dL | FPG 80-110 mg/dL
Number analyzed (Participants) | 112 | 112
percentage of participants | 41.1 | 26.8
Statistical Analysis 1: Comparison: FPG 70-90 mg/dL vs FPG 80-110 mg/dL; Test type: Non-Inferiority or Equivalence — The hypothesis was that there would be no difference in efficacy as measured by the proportion of subjects reaching HbA1c level <= 6.5% between the two FPG titration arms (70-90 mg/dL and 80-110 mg/dL, respectively) with a non-inferiority margin of 20%. If non-inferiority of the 70-90mg/dL arm was established, superiority was to be tested using a Logistic regression model with baseline HbA1c as a covariate. Superiority was to be concluded if the odds ratio was significantly greater than 1; p = 0.0064, Regression, Logistic; Odds Ratio (OR) = 2.34, 95% CI [1.27 to 4.30]

3. Secondary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c) Percentage From Baseline
Description: Change in glycosylated haemoglobin A1c (HbA1c) percentage from baseline measured from week -2 to week 20
Time Frame: week -2, week 20
Population: The intent-to-treat (ITT), LOCF (last observation carried forward) population. One Subject in 70-90 group, however, had a missing baseline value, therefore, no change from baseline could be calculated.
Measure: Least Squares Mean (Standard Error); unit: percentage point change
Arm/Group | FPG 70-90 mg/dL | FPG 80-110 mg/dL
Number analyzed (Participants) | 111 | 112
percentage point change | -1.229 (0.061) | -0.958 (0.061)
Statistical Analysis 1: Comparison: FPG 70-90 mg/dL vs FPG 80-110 mg/dL; Test type: Superiority or Other; p = 0.0019, ANCOVA; The analyses for HbA1c were adjusted for baseline HbA1c values; LSMean = -0.271, 95% CI [-0.441 to -0.101]

4. Secondary Outcome: Incidence of Hypoglycaemic Episodes (All, Major, Minor and Symptoms Only)
Description: Incidence of hypoglycaemic episodes (all, major, minor and symptoms only) occurring during the treatment period from week 0 to week 20. Classification was as follows:
  * If subject was unable to treat himself: Major incidence.
  * If subject could treat himself and plasma glucose was less than 3.1 mmol/l: Minor incidence.
  * If subject could treat himself and plasma glucose was equal to or greater than 3.1 mmol/l, or there was no plasma glucose measurement: Symptoms only.
Time Frame: weeks 0-20
Population: The safety population consists of all subjects exposed to study drug.
Measure: Number; unit: number of events
Arm/Group | FPG 70-90 mg/dL | FPG 80-110 mg/dL
Number analyzed (Participants) | 121 | 122
number of events
  All | 333 | 227
  Major | 1 | 0
  Minor | 225 | 136
  Symptoms only | 107 | 91

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a time span of 20 weeks.
Description: The safety population (safety analysis set) contained all subjects who took at least one dose of study medication.
Arm/Group | FPG 70-90 mg/dL | FPG 80-110 mg/dL
Serious Adverse Events (participants affected / at risk) | 5/121 | 4/122
Other Adverse Events (participants affected / at risk) | 45/121 | 30/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FPG 70-90 mg/dL (N=121) | FPG 80-110 mg/dL (N=122)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FPG 70-90 mg/dL (N=121) | FPG 80-110 mg/dL (N=122)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.